CLINICAL TRIAL: NCT00666016
Title: Double-Blind vs Placebo, Randomized, Exploratory Study to Assess the Short Term Effect on Liver Enzymes and the Safety of TRO19622 500 mg QD for One Month in Patients With Non-Alcoholic Steatohepatitis (NASH)
Brief Title: Exploratory Study to Assess the Short Term Effect on Liver Enzymes and the Safety of TRO19622 in Patients With Non-Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Trophos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN29850; TRO19622 CL E Q 1159-1 (Other: trophos id)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH)
Keywords: non alcoholic steatohepatitis nash hepatoprotective hepatoprotection ALT AST new drug candidate interventional study TRO19622 Trophos cholest-4-en-3-one oxime
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — olesoxime

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRO19622 (Experimental): TRO19622 500 mg
  Interventions: Drug: TRO19622
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRO19622 — TRO19622 500 mg once a day before noon meal during 6 weeks
  Other Names: Olesoxime
  Arms: TRO19622
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, the tolerability and the short term effect on liver enzymes of TRO19622 500 mg for one month in patients with Non-Alcoholic Steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects older than 18 years.
* Persistent ALT elevation (> 2 times the ULN of the local laboratory of the investigating site) over 6 months prior to entry into study.

  * No more than one ALT value within the normal range in the past year.
  * Patients must have had an ALT measurement at least once every 6 months within the year before inclusion.
* Histologically confirmed diagnosis of steatohepatitis on biopsy within 2 years prior to entry into protocol.
* Compensated liver disease with the following hematologic, biochemical, and serological criteria on entry into protocol:

  * Hemoglobin > 11 gm/dL for females and > 12 gm/dL for males
  * White blood cell (WBC) > 2.5 K/UL
  * Neutrophil count > 1.5 K/UL
  * Platelets > 100 K/UL
  * Total bilirubin < 35 µmol/L)
  * Albumin > 36 g/L
  * TP > 80% .
  * Serum creatinine within normal limits
* No other cause of chronic liver disease (autoimmune,primary biliary cirrhosis, HBV, Wilson, alpha-1-antitrypsin deficit, hemochromatosis etc\dots )
* If applicable, have a stable diabetes, defined as HbA1c < 9% and fasting glycemia < 10 mmol/L,no changes in medication in the previous 6 months, and no new symptoms associated with diabetes in the previous 3 months.
* If applicable have a stable metabolic condition (diagnosis made at least 6 months before inclusion), without major weight or laboratory tests changes.
* Negative pregnancy test or post menopausal.
* Have an electrocardiogram (ECG) without any clinically significant abnormality.
* Subjects must be willing to give written informed consent.

Exclusion Criteria:

* Evidence of another form of liver disease.
* History of excess alcohol ingestion: daily alcohol consumption >30 g/day (3 drinks per day) for males and >20 g/day (2 drinks/day) for females.
* Unstable metabolic condition: Weight change > +/- 10% in the previous year, diabetes with poor glycemic control (HbA1c >9%),introduction of an antidiabetic or of an anti-obesity drug in the past 6 months prior to screening.
* History of gastrointestinal bypass surgery or ingestion of drugs known to produce hepatic steatosis including corticosteroids,high-dose estrogens, methotrexate, tetracycline or amiodarone in the previous 6 months.
* Significant systemic or major illnesses other than liver disease,including congestive heart failure, coronary artery disease, cerebrovascular disease, pulmonary disease, renal failure, organ transplantation, serious psychiatric disease,malignancy that, in the opinion of the investigator would preclude treatment with TRO19622 and/or adequate follow up.
* HIV infection.
* Active substance abuse, such as inhaled or injection drugs within the previous year.
* Pregnancy or inability to practice adequate contraception in women of child-bearing potential.
* Active malignancy except cutaneous basocellular carcinoma.
* Any other condition which, in the opinion of the investigator would impede competence or compliance or possibly hinder completion of the study.
* Body mass index (BMI) >40 kg/m2 (obesity Grade III).
* Type 1 diabetes or Insulin-treated type 2 diabetes.
* Hemostasis disorders or current treatment with anticoagulants.
* History of, or current cardiac dysrhythmias and / or a history of cardiovascular disease, including myocardial infarction, except patients with only well controlled hypertension.
* Participation in any other investigational drug or therapy study within the previous 3 months.
* Be possibly dependent on the Investigator or the Sponsor (eg, including, but not limited to, affiliated employee).
* Medications that could interfere with TRO19622 absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-04-15 (Actual); Primary Completion 2009-02-05 (Actual); Study Completion 2009-02-05 (Actual)

PRIMARY OUTCOMES:
Mean change in ALT as assessed by an ANCOVA with the following covariates: treatment, gender, subject and time and a non parametric test (Conover-Salsburg). | Mean change in ALT at V1 (Day15) and V2 (Day 30)

SECONDARY OUTCOMES:
Sustained reduction in ALT to either 50% of baseline or value < or equal to ULN. Sustained reduction serum AST and GGT.Clinical and laboratory safety. | V1 (Day 15), V2 (Day 30) and V3 (Day 60)

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Ratziu, MD, Principal Investigator — GH PITIE-SALPETRIERE
Locations (5):
- France (5):
  - CHU AMIENS, Service d'Hépato-Gastroentérologie, Amiens
  - Centre Hospitalier de Hyères, Hôpital de Jour, Service d'Hépato-Gastro-Entérologie, Hyères
  - Hôpital Saint Joseph, Service d'Hépato-Gastro-Entérologie, Marseille
  - Hôpital Archet 2 - Pôle de Référence Hépatite C (Niveau -2) - 151, route Saint Antoine de Ginestière, Nice
  - Groupe Hospitalier Pitié-Salpétrière - Sce Hépato-Gastroentérologie - 47-83 Bd de l'Hôpital, Paris